CLINICAL TRIAL: NCT03147872
Title: Lo2 Phase II: A Comparison of Live Birth Rates Between Embryos Cultured in 2% vs. 5% After Day 3 of Embryo Culture
Brief Title: Evaluation of the Impact of Reduced Oxygen Concentration on Live Birth Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Collaborators: Instituto Universitario IVI (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RMA-2017-02
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients and care providers will be masked as to which embryo is randomized to each condition. Investigators will be masked until the data are analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5% Oxygen (No Intervention): All patients' embryos will be cultured in 5% oxygen from day 1 through 3 of development. After day 3 of development, patients randomized to this arm will continue to have their embryos cultured at 5% oxygen until they are deemed to be clinically usable or not clinically usable (as per standard protocol).
- 2% Oxygen (Experimental): All patients' embryos will be cultured in 5% oxygen from day 1 through 3 of development. After day 3 of development, patients randomized to this arm will have their embryos cultured at 2% oxygen until they are deemed to be clinically usable or not clinically usable (per standard criteria).
  Interventions: Other: 2% Oxygen

INTERVENTIONS:
Other: 2% Oxygen — 2% oxygen concentration in the incubator in which embryos are being cultured after day 3 of development
  Arms: 2% Oxygen

SUMMARY:
Clinical in vitro fertilization relies on successful embryo culture. The primary goal of embryo culture is to attempt to recapitulate the in vivo conditions as much as possible. In the past decade, the majority embryo culture has been performed at 5% oxygen due to the discovery that the oxygen tension in the fallopian tube (where the embryo is located for the first 3 days after fertilization) is 5%. However, relatively recent studies have demonstrated that the oxygen tension in the uterus (where the embryo is located after day 3) is closer to 2%. This study is a randomized controlled trial that will compare pregnancy rates between embryos cultured in 2% versus 5% after day 3 of development.

DETAILED DESCRIPTION:
Significant progress has been made in characterizing the optimal environment for a developing embryo in culture. These efforts have been based on the premise that clinical embryo culture should mimic the in vivo environment. To this end, investigators have gone to great lengths to recreate every aspect of the natural setting to which the early embryo is exposed. This focused approach has led to significant modifications of the embryo culture system in the modern in vitro fertilization (IVF) lab and ultimately to improvements in pregnancy rates.

One area that has been subject to significant scrutiny is the relationship between incubator oxygen concentration and early embryonic development. Oxygen plays a central role in embryonic metabolism. The mechanism governing its utilization is dependent on the stage of embryonic development. During the first 3 days of development, oxygen reaches the embryo via passive diffusion and its concentration gradient is regulated by oxygen consumption during oxidative phosphorylation. Inefficiencies in this process - due to compromised integrity of the inner mitochondrial membrane or alterations in substrate availability - can result in excessive production of harmful reactive oxygen species which can cause significant damage to cellular machinery and ultimately lead to embryonic arrest.

The concentration of oxygen that the embryo in culture is exposed to can also impact this delicately balanced system and alter the metabolic health of an embryo. Historically, atmospheric oxygen concentration (approximately 20%) was exclusively used in human IVF laboratories for embryo culture. However, multiple investigations subsequently found that the physiologic concentration of oxygen within the female reproductive tract is well below atmospheric levels, being consistently measured at <10%. These observations led to multiple trials comparing atmospheric oxygen concentrations to 5% oxygen in embryo culture. These studies demonstrated significant perturbations in gene expression, protein secretion, and suboptimal utilization of amino acids and carbohydrates in embryos cultured in atmospheric oxygen. The same comparisons were made in clinical IVF studies and demonstrated that embryos cultured in 5% oxygen consistently resulted in an increase in clinical pregnancy rate and live birth rate. A meta-analysis of this topic suggested that a clinic with a baseline live birth rate of 30% could expect an improvement as great as 13% when culturing embryos at 5% O2.

As a result of these compelling data, most modern IVF programs now exclusively culture embryos at 5% oxygen concentration. However, some have proposed that the oxygen concentration to which the embryo is exposed after day 3 of development is actually lower than 5%. These data originate from the idea that the embryo crosses the utero-tubal junction on day 3 of development in vivo. Multiple studies have demonstrated that the oxygen concentration in the uterus is actually lower than that in the fallopian tube at approximately 2%. Thus, the most physiologic embryo culture system would culture embryos in 5% oxygen until day 3 and then decrease the oxygen concentration to 2% until transfer or cryopreservation on day 5 or 6.

A change in the optimal oxygen concentration for an embryo on day 3 would fit with a general shift in metabolic requirements of embryos seen at this stage of development. Activation of the embryonic genome occurs on day 3 which prompts a significant increase in biosynthetic activity. The metabolic behavior of embryos also shifts substantially during this time. The embryo changes its metabolic strategy from oxidative phosphorylation to glucose based metabolism in the form of the aerobic glycolysis and the citric acid cycle. During this process, termed compaction, embryos exhibit greatly increased oxygen consumption.

The physiologic environment of the female reproductive tract tends to mirror the metabolic needs of the developing preimplantation embryo. As the embryo shifts its metabolic strategy after compaction and upon entering the uterus, it is certainly possible that a reduced oxygen concentration in the uterus may best support the energy producing mechanisms of this stage in embryonic development. Recapitulating this environment in culture may enhance embryonic development and long term health of pregnancies resulting from IVF.

This theory has been corroborated in two recent pilot studies. The first study, recently awarded the Prize Paper Award at the 2016 American Society for Reproductive Medicine Scientific Meeting, randomized embryos donated to research to 2% or 5% oxygen concentration after day 3 of development and found that embryos were twice as likely to blastulate if they were cultured in 2% oxygen concentration. However, embryos studied in this investigation were either abnormally fertilized or warmed from cryopreservation on day 3 after being donated to research. None were intended for clinical use.

With these limitations in mind, our group has recently completed a study utilizing embryos intended for clinical use (Copernicus IRB: RMA-2016-02). In this study, we enrolled 60 patients and split all ongoing embryos on day 3 of development to culture in either 2% or 5% oxygen until the blastocyst stage. The results have not yet been published, but culture in 2% oxygen after day 3 produced more blastocysts than culture in 5% oxygen. In total, 30 patients had more embryos reach blastocyst in 2% oxygen, while only 17 patients had more embryos reach blastocyst in 5% oxygen. Ten patients had an equal number in both conditions (3 withdrew from the study). This difference reached statistical significance.

This initial study was designed to specifically evaluate the developmental performance of embryos in both conditions. However, there are also some pregnancy data available from those patients who have proceeded to transfer these embryos. In this initial study, culture conditions had no impact on the decision of which embryo to transfer. This was blinded to embryologists and patients and only typical morphology criteria were utilized. Again, of patients who have proceeded to embryo transfer, embryos that had been cultured in 2% oxygen have performed better than those exclusively in 5% (88.9% [16/18] vs. 62.5% [15/24]

However, this initial study was not designed to specifically test the question of whether 2% versus 5% oxygen in extended culture produces better pregnancy outcomes. The patients were not randomized to either 2% or 5% oxygen. Thus, current pregnancy data is prone to some bias and a better controlled study is needed evaluate the impact of reduced oxygen concentration in culture on the most important outcomes: live birth rate.

Purpose of Proposed Study This study seeks to compare clinical outcomes of embryos cultured at 2% oxygen concentration and 5% oxygen concentration after compaction. The primary outcome under study will be live birth rate. Secondary outcomes will include miscarriage rate, gestational age at delivery, birth weight at delivery, embryo blastulation rate, embryo ploidy status (aneuploid or euploid) and morphologic parameters (expansion, inner cell mass grade, trophectoderm grade). The cumulative live birth rate of all embryos that originate from the study stimulation cycle will also be collected and analyzed. This will theoretically reveal whether any advantage in the number of available blastocysts for transfer translates to greater reproductive efficiency when extended culture is performed at 2% oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Anti-mullerian hormone level (AMH) > 1.0 ng/mL
* Must have at least one surviving embryo on day three of development
* Male partner with >100,000 total motile spermatozoa per ejaculate (donor sperm acceptable)
* Body Mass Index < 35

Exclusion Criteria:

* Diagnosis of endometrial insufficiency, as defined by prior cycle with maximal endometrial thickness <6mm, abnormal endometrial pattern (failure to attain a trilaminar appearance), or persistent endometrial fluid
* Use of oocyte donation
* Use of gestational carrier
* Use of sperm obtained via surgical procedure
* Presence of hydrosalpinges that communicate with endometrial cavity
* Single gene disorders, chromosomal translocations or any other disorders requiring more detailed embryo genetic analysis
* Couples seeking gender selection for family balancing
* Completion of the protocol requires a single embryo transfer of an embryo as part of the study. Thus, patients pursuing embryo banking cycles will be excluded from the study.
* Double embryo transfer

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Genotypically female (with functioning ovaries)
Enrollment: 280 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Live Birth Rate | through study completion, an average of 1 year
  Delivery of a fetus after 20 weeks of gestation (WHO definition)

SECONDARY OUTCOMES:
Miscarriage Rate | through study completion, an average of 1 year
  Number of pregnancy losses after visualization of a gestational sac and yolk sac on ultrasound
Gestational Age at delivery | through study completion, an average of 1 year
  The number of weeks gestation completed prior to delivery of the fetus
Birthweight at delivery | through study completion, an average of 1 year
  Weight in grams of fetus at time of delivery
Embryo blastulation rate | through study completion, an average of 1 year
  Number of embryos that progress to the blastocyst developmental stage per fertilized ova
Embryo ploidy status | through study completion, an average of 1 year
  The percentage of embryos that are deemed euploidy by preimplantation genetic screening
Embryo morphologic parameters | through study completion, an average of 1 year
  Assignment of morphologic grade of embryos (as per modified Gardner's criteria)
Cumulative live birth rate | through study completion, an average of 1 year
  The number of live births (per definition above) achieved from all embryos derived from the in vitro fertilization cycle involved in the study for a given patient

CONTACTS AND LOCATIONS:
Overall Officials: Scott Morin, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey; Daniel J Kaser, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fischer B, Bavister BD. Oxygen tension in the oviduct and uterus of rhesus monkeys, hamsters and rabbits. J Reprod Fertil. 1993 Nov;99(2):673-9. doi: 10.1530/jrf.0.0990673. PMID 8107053
- [Background] Bontekoe S, Mantikou E, van Wely M, Seshadri S, Repping S, Mastenbroek S. Low oxygen concentrations for embryo culture in assisted reproductive technologies. Cochrane Database Syst Rev. 2012 Jul 11;2012(7):CD008950. doi: 10.1002/14651858.CD008950.pub2. PMID 22786519
- [Background] Gardner DK, Wale PL. Analysis of metabolism to select viable human embryos for transfer. Fertil Steril. 2013 Mar 15;99(4):1062-72. doi: 10.1016/j.fertnstert.2012.12.004. Epub 2013 Jan 8. PMID 23312219
- [Background] Rinaudo PF, Giritharan G, Talbi S, Dobson AT, Schultz RM. Effects of oxygen tension on gene expression in preimplantation mouse embryos. Fertil Steril. 2006 Oct;86(4 Suppl):1252-65, 1265.e1-36. doi: 10.1016/j.fertnstert.2006.05.017. PMID 17008149
- [Background] Meintjes M, Chantilis SJ, Douglas JD, Rodriguez AJ, Guerami AR, Bookout DM, Barnett BD, Madden JD. A controlled randomized trial evaluating the effect of lowered incubator oxygen tension on live births in a predominantly blastocyst transfer program. Hum Reprod. 2009 Feb;24(2):300-7. doi: 10.1093/humrep/den368. Epub 2008 Oct 16. PMID 18927130